CLINICAL TRIAL: NCT01206933
Title: The Effect of HIV Tat Protein on HCV Replication in an In-vitro Model System.
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: GWUIRB #061012
Record Dates: First submitted 2010-09-17; First posted 2010-09-22 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2010-09

CONDITIONS: Human Immunodeficiency Virus (HIV); Hepatitis C, Chronic
Keywords: HIV/HCV Coinfection; Tat Protein; HCV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Detectable HIV RNA and HCV RNA: HIV and HCV co-infected with detectable HIV RNA and HCV RNA
- Undetectable HIV and Detectable HCV: HIV and HCV infected, HIV RNA Undetectable(treated) and Detectable HCV RNA.
- Undetectable HIV and HCV: HIV and HCV infected, Undetectable HIV RNA and HCV RNA
- Undetectable HCV: HCV(mono-infected,) HCV RNA undetectable
- Detectable HCV RNA: Monoinfected HCV, detectable RNA
- Detectable HIV RNA: Monoinfected HIV, Detectable RNA

SUMMARY:
Investigators in the Division of Infectious Diseases and the Departments of Biochemistry and Molecular Biology of The George Washington University Medical Center are carrying out a research study to determine why patients with Human Immunodeficiency Virus (HIV) and Hepatitis C virus (HCV) co-infection (HIV/HCV) have a more rapid and progressive course of HCV infection, leading to fatty infiltration of the liver and cirrhosis.

DETAILED DESCRIPTION:
Samples will be collected from 4 groups of patients with HIV/HCV infection, identified by the virologic control of either HIV, HCV, or both. Sera will be used in an in-vitro hepatocyte model of hepatitis C infection to better understand the pathogenesis of HIV/HCV co-infection, and to gain insight into intracellular mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following criteria:

  1. detectable HIV RNA and detectable HCV RNA
  2. undetectable HIV RNA (treated) and detectable HCV RNA
  3. undetectable HIV RNA (treated) and undetectable HCV RNA
  4. undetectable HCV RNA (mono-infected)
  5. detectable HCV RNA (mono-infected)
  6. detectable HIV RNA (mono-infected)

Participants will be men and women, ages 18 and older, and who are patients being seen in the clinics of the Medical Faculty Associates, and meet the above criteria.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four groups of subjects will be included in this study, with 5 participants in each group:
  1. detectable HIV RNA (Ribonucleic Acid) and detectable HCV RNA
  2. undetectable HIV RNA (treated) and detectable HCV RNA
  3. undetectable HIV RNA (treated) and undetectable HCV RNA
  4. undetectable HCV RNA (mono-infected)
  5. detectable HCV RNA (mono-infected)
  6. detectable HIV RNA (mono-infected)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Laboratory analysis of Tat Protein | Single sample analysis
  The validation that HIV Tat protein is a potent inducer of HCV in dual infected patients will likely lead to anti-tat therapy to manage HCV patients for whom treatment options are rather limited.

CONTACTS AND LOCATIONS:
Overall Officials: David Parenti, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No